CLINICAL TRIAL: NCT02304952
Title: Eccentric Exercise or Radiofrequent Microtenotomy as Treatment of Chronic Lateral Epicondylalgia - a Randomized Controlled Trial
Brief Title: Eccentric Exercise or Radiofrequent Microtenotomy as Treatment of Lateral Epicondylalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capio Sankt Görans Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lateral epicondylalgia
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Tennis Elbow
Keywords: Lateral epicondylalgia; Pain; Function; Physiotherapy; Quality of Life
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric exercise (Active Comparator): Conservative treatment with eccentric exercise as self-training
  Interventions: Other: Eccentric exercise
- Radiofrequency microtenotomy (Active Comparator): A minimally invasive surgery (Topaz) and eccentric exercise as postoperative treatment
  Interventions: Procedure: Radiofrequency microtenotomy; Device: Arthrocare Topaz MicroDebrider

INTERVENTIONS:
Procedure: Radiofrequency microtenotomy — For the minimally invasive surgery will Arthrocare Topaz MicroDebrider device be used. A small incision will be made and the tip of the device is placed on surface of the tendon to structure and activated for 0.5 second, at 5 mm distance intervals on the tendon creating a grid-like pattern.
  Other Names: Minimally invasive surgery
  Arms: Radiofrequency microtenotomy
Other: Eccentric exercise — Eccentric exercise for 3 months. The exercise will be performed once a day with 3 set and 5 reps, women start with 0.5 and men 1.0 kilo with a 10 % increase every week.
  Arms: Eccentric exercise
Device: Arthrocare Topaz MicroDebrider
  Arms: Radiofrequency microtenotomy

SUMMARY:
The aim is to study the effects related to function and pain during eccentric exercise and surgery with radiofrequency microtenotomy as post-surgical rehabilitation, compared with only eccentric exercise, in patients with lateral epicondylalgia unilaterally.

DETAILED DESCRIPTION:
Of those affected by lateral epicondylalgia will 90% be free of symptoms within 8 months to 2 years with conservative treatment. In this study surgical radiofrequency microtenotomy and eccentric exercise for chronic (more than two year) lateral epicondylalgia that is unilaterally will be used as treatment. Patients is randomized to a group with eccentric exercise or a group with surgical radiofrequency microtenotomy and postoperatively eccentric exercise. Home based eccentric exercise program is instructed by a physical therapist and is performed for three months. Women start with 0.5 kg and men 1.0 kg weight, they perform 3 sets with 5 reps once a day and register pain and exercise in a diary. Function, pain and quality of life will be followed and are carried out after 6 weeks and after 3, 6 and 12 months. The surgery and eccentric exercise is instructed and followed at the investigators clinic.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 and under the age of 70 year
* lateral epicondylalgia at least two year
* tried conservative treatment

Exclusion Criteria:

* complicated systemic diseases (such as diabetes)
* understand spoken and or/written instructions in Swedish

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Function. | 12 month
  Function measured with the DASH (Disability of Arm-Shoulder-Hand) Questionnaire and Jamar dynamometer as static maximum grip strength.
Pain. | 12 month
  Pain estimated with Visual Analogue Scale (VAS 0-100 mm).

SECONDARY OUTCOMES:
Quality of life. | 12 month
  The Short Form-12 (SF-12) is a questionnaire which measures Quality of Life (QoL), which are both physically and emotionally based.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Heijne, PT, PhD, Study Director — Karolinska Institutet
Locations (1):
- Capio Sankt Göran Hospital, Stockholm, Stockholm County, Sweden